CLINICAL TRIAL: NCT05249777
Title: A Phase III, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of TD0069 Capsule for Patients With Mild to Moderate COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: CLINICAL RESEARCH VIET NAM SKILL TRAINING AND CONSULTING COMPANY LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TD0069-COVID19-III
Record Dates: First submitted 2022-02-21; First posted 2022-02-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Study subjects are randomized in a 2:1 ratio to 14 days treatment with TD0069 (3 capsules x 3 times/day) or Placebo (3 capsules x 3 times/day) based on a randomization block size of 6.
Who Masked: Participant, Investigator
Masking Description: Blinding is performed by the same appearance of TD0069 and placebo. The request for unblinding is done in accordance with the study protocol in cases of SAEs with the request of the investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TD0069 (Experimental): Standard dose, 3 capsules/time x 3 times/day x 14 days before breakfast, lunch, and dinner combined with standard treatment.
  Interventions: Drug: TD0069 hard capsule
- Placebo (Placebo Comparator): Standard dose, 3 capsules/time x 3 times/day x 14 days before breakfast, lunch, and dinner combined with standard treatment
  Interventions: Drug: TD0069 Placebo

INTERVENTIONS:
Drug: TD0069 hard capsule — TD0069 hard capsule (800 ± 7.5% mg/capsule) contains 600 mg fine powder of mixed herbal medicines and 200 mg excipients.
  Other Names: Sunkovir
  Arms: TD0069
Drug: TD0069 Placebo — TD0069 placebo (800 ± 7.5% mg/capsule) contains excipients
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The acute pneumonia pandemic caused by a new strain of corona virus 2019, namely as COVID-19 by the World Health Organization (WHO), is a pandemic caused by SARS-CoV-2 virus. The reported symptoms vary from fever or chills, cough, shortness of breath, to muscle aches, headaches, loss of taste or smell.

The capsule TD0069 is a product based on the traditional medicine named "Ren shen bai du san" which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

DETAILED DESCRIPTION:
The acute pneumonia pandemic caused by a new strain of corona virus 2019, namely as COVID-19 by the World Health Organization (WHO), is a pandemic caused by SARS-CoV-2 virus. The reported symptoms have included, but are not limited to fever or chills, cough, shortness of breath, muscle aches, headaches, loss of taste or smell, diarrhea, dizziness, sore throat, abdominal pain, anorexia, and vomiting.

The capsule TD0069 is a product based on the traditional prescription named "Ren shen bai du san" which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

The study compares between standard dose regimen of TD0069 combined with standard treatment in COVID-19 patients and only standard treatment in COVID-19 patients. A sample size of 570 patients, 380 in TD0069 arm and 190 in Placebo arm.

All participants will be treated and followed up in 14-day period. In case the participant meets the discharge criteria before 14 days, discontinuing the study drug will be done at the discretion of the investigators.

Firstly, screening procedures occur at Day 1. Secondly, periodic assessments are conducted daily from Day 2-14. Finally, end-of-study assessments are conducted according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Human, age ranged from 18 to 65 years old, Vietnamese nationality.
* Confirmed diagnosis with a positive test for SARS-CoV-2 by real-time RT-PCR.
* Patients with mild and moderate Covid-19 disease according to the classification of clinical severity of SARS CoV2 of the Ministry of Health (No. 4689/QĐ-BYT Decision dated October 6, 2021 of the Ministry of Health about promulgating guidelines for diagnosis and treatment Covid-19 ): patient is awake, breathing rate ≤ 25 times/min, SpO2 ≥ 94% when breathing room air, and may have difficulty breathing when exertion.
* Provision of signed informed consent.
* Being able to comply with study procedures and treatment, in the opinion of the investigator.
* Patients with at least 01 of 11 main symtoms of Covid-19

Exclusion Criteria:

* Symptoms of severe upper and lower respiratory tract infections (as defined by WHO)1 such as dyspnea, SpO2 < 94%.
* Patients with acute respiratory distress in any of the following groups:

  * Respiratory failure due to hypoxemia when PaO2 was less than 60mmHg with room air.
  * Respiratory failure due to hypercapnia when PaCO2 was above 50mmHg.
  * Mixed respiratory failure due to the combination of hypoxemia and hypercapnia.
* Allergy/intolerance to any ingredient of the investigational products.
* Patients who are not able to orally use the investigational products.
* Patients who have been treated with corticoid at the screening.
* Participants who were not able to comply with study procedures and treatment, in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
The rate of patients with serious diseases/conditions related to Covid-19 | up to 28 days
  Severe progression within 28 days of randomization, including occurrence of any 1 of the following events: Acute respiratory distress syndrome (ARDS) with high-flow nasal cannula oxygen therapy (HFNC) and invasive mechanical ventilation therapy, sepsis, septic shock , multiple organ failure requiring intensive care (ICU), other critical conditions, and death
Daily symptoms improvement | up to 14 days
  Symptom severity was assessed in accordance with the Covid-19 symptom assessment questionnaire of National Early Warning Score. The higher patient's score, the more severe symtoms.
Time to clinical symptom resolution | up to 14 days
  Mean time from randomization to symptom resolution in terms of general, cardiovascular, respiratory, digestive, musculoskeletal, neurological, and dermatological symptoms
The rate and severity grade of adverse events related to the investigational product | up to 28 days
  Absolute number of immediate adverse events classified by severity level Percentages were calculated as the total number of immediate adverse events classified by severity level divided by the total number of subjects.

SECONDARY OUTCOMES:
The rate of Covid-19 diseases according to traditional medicine | up to 14 days
  Covid-19 diseases according to traditional medicine
Time to symptom resolution of Covid-19 diseases according to traditional medicine | up to 14 days
  Mean time from randomization to symptom resolution of Covid-19 diseases according to traditional medicine
The length of hospital stay | up to 14 days
  Date of discharge minus date of admission
The rate of Number of Participants Until First Non-detectable SARS-CoV-2 in Nasopharyngeal (NP) Swabs | Day 5, day 7, day 9, and day 14
  The proportion of participants until first non-detectable SARS-CoV-2 in nasopharyngeal (NP) swabs will be estimated for each randomized arm (drug versus placebo) at day 5, day 9, day 14 after randomization.
The quality of life at day 0, day 7, day 14, and day 28 | Day 0, day 7, day 14, and day 28
  Quality of life score accordance with EQ-5D-5L questionnaire table

CONTACTS AND LOCATIONS:
Overall Officials: Loc Huynh Nguyen, SL II., MD., Principal Investigator — Traditional Medicine Institute in Ho Chi Minh City; Lan Truong Thi Ngoc, PhD., MD., Principal Investigator — Traditional Medicine Institute in Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - Traditional Medicine Institute in Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh
  - Hanoi Hospital of Traditional Medicine, Hà Nội